CLINICAL TRIAL: NCT00580944
Title: Combined Alexandrite and Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participant enrolled
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20064992
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
Keywords: Port wine stain; progressive malformation of human skin
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Port Wien Stain Birthmark (Experimental): Combined alexandrite and pulsed dye laser treatment of port wine stain birthmarks
  Interventions: Procedure: laser treatment of port wine stain birthmarks

INTERVENTIONS:
Procedure: laser treatment of port wine stain birthmarks — Combined alexandrite and pulsed dye laser treatment of port wine stain birthmarks

SUMMARY:
Port wine stain is a congenital, progressive vascular malformation of skin involving post-capillary venules that occurs in an estimated 4 children per 1,000 live births. Approximately 1,200,000 individuals in the United States and twenty-six million people worldwide have Port wine stain birthmarks.

Since most of the malformations occur on the face, Port wine stain is a clinically significant problem in the majority of patients. Port wine stain should not be considered a cosmetic problem but a disease with potentially devastating psychological and physical complications. Personality development is adversely influenced in virtually all patients by the negative reaction of others to a "marked" person. Port wine stain are initially flat red macules, but lesions tend to darken progressively to purple, and by middle age, often become raised as a result of the development of vascular nodules. Hypertrophy of underlying soft tissue further disfigures the facial features of many patients.

DETAILED DESCRIPTION:
The researcher can use alexandrite and pulsed dye lasers pulses combined delivery to improve port wine stain blanching. The alexandrite and pulsed dye lasers are both approved by the Food and Drug Administration for the treatment of Port wine stain. However, the degree of port wine stain blanching seen following either alexandrite or pulsed dye lasers treatment remains variable and unpredictable. Treatment of port wine stains can use either alexandrite or pulsed dye alone and with the combined delivery of alexandrite and pulsed dye lasers pulses.

ELIGIBILITY:
Inclusion Criteria:

* Port Wine Stain suitable for comparison testing
* Age > 12 years and older
* minor will be accompanied by parents or guardians during laser treatment
* Apparent good health as documented by medical history

Exclusion Criteria:

* History of photodermatoses or skin cancer
* Any therapy within the previous two months to the proposed Port Wine Stain treatment sites
* Current participation in any other investigational drug or device evaluation
* Concurrent use of known photosensitizing drugs

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Port Wine Stain Birthmarks blanching | 8 weeks
  Post-treatment blanching responses can determine quantitatively by visual reflectance spectroscopy and compare with pre-treatment measurements of Port Wine Stain fractional blood volume

CONTACTS AND LOCATIONS:
Overall Officials: JOHN S NELSON, M.D,Ph.D, Principal Investigator — Beckman Laser Institute